CLINICAL TRIAL: NCT06680986
Title: Echocardiographic Analysis by Artificial Intelligence in Hypertension
Acronym: CARDINAL
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0643; 898 (Other: HCL)
Record Dates: First submitted 2024-01-22; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Arterial Hypertension
Keywords: Hypertension; HTN; Arterial Hypertension; Artificial Intelligence; AI; Cardiac remodelling; Left ventricular hypertrophy
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — Arterial Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hypertensive patients: Patients having undergone a blood pressure assessment during hospitalization in the Fédération de Cardiologie at Hôpital de la Croix Rousse and Hôpital Lyon Sud from January 2018 to December 2021
  Interventions: Other: Clinical cardiac parameters (Arterial pressure, number of anti-hypertensive medications, and the NT-proBNP measurements)

INTERVENTIONS:
Other: Clinical cardiac parameters (Arterial pressure, number of anti-hypertensive medications, and the NT-proBNP measurements) — The degree of severity of the hypertension will have been previously diagnosed for each patient with the help of the blood pressure measurements, the number of antihypertensive treatments and the NT-proBNP measurement which is correlated with the left intraventricular pressure and the mass of the left ventricle. This information will be used (i) to guide the structuring of the pathology representation space during the learning phase from a sub-population (a portion of the collected database that will be used for training algorithms); (ii) to serve as an endpoint from a test sub-population (the remaining portion of the database collected).

SUMMARY:
The objective of this study is to develop artificial intelligence (AI) tools to characterize cardiac remodelling in arterial hypertension through the analysis of routine imaging data (echocardiography) coupled with patient data. More precisely, this study will make it possible (i) to represent in a relevant way the spectrum of the cardiac repercussions of a population affected by hypertension to better characterize the progress of the pathology, in particular vis-à-vis the more ambiguous subjects to be characterized ("grey" area); (ii) to develop tools for the automatic quantification of cardiac function (segmentation and robust monitoring of the myocardium during the cardiac cycle, for the dynamic analysis of the shape and global deformation of the heart) and therefore to extract descriptors richer in cardiac function than those currently used in clinical routine.

ELIGIBILITY:
Inclusion Criteria Patients who underwent a comprehensive blood pressure assessment during hospitalization in the Cardiologic Federation at Croix Rousse Hospital and Lyon Sud Hospital between January 2018 and December 2021.

Exclusion Criteria Patients who are minors. Patients under curatorship or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a comprehensive hypertension assessment during hospitalization in the Cardiologic Federation at Croix Rousse Hospital and Lyon Sud Hospital between January 2018 and December 2021
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Arterial Blood Pressure | Baseline
  This measure will assess the arterial blood pressure in millimeters of mercury (mmHg). Blood pressure measurements will include both systolic and diastolic values. This measurement will be used to evaluate the severity of hypertension and track changes over the course of the study.
Number of Antihypertensive Medications | Baseline
  This measure will record the number of antihypertensive medications prescribed to each patient. The data will be used to assess the intensity of the treatment regimen required to control blood pressure levels in participants.
  Unit of Measure: Count of medications (integer)
NT-proBNP Concentration | Baseline
  This measure will assess plasma concentrations of N-terminal pro b-type natriuretic peptide (NT-proBNP), a biomarker correlated with left ventricular pressure and mass. NT-proBNP levels will be analyzed in picograms per milliliter (pg/mL) to evaluate cardiac stress associated with hypertension.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: Undecided